CLINICAL TRIAL: NCT04112940
Title: Physiological Flow of Liquids in Head and Neck Cancer Patients: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-5190; 5R01DC011020 (NIH); CAPCR 16-5190 (NIH_HNC) (Other: UHN Research Ethics Board)
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Deglutition Disorders; Oropharynx Cancer
Keywords: Swallowing
MeSH Terms: conditions — Deglutition Disorders; Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with oropharyngeal cancer: Adult participants who have completed radiation therapy for oropharyngeal cancer within the past 3 months will undergo a swallowing x-ray study in which they will swallow up to 15 liquid stimuli prepared to different consistencies using starch and gum based thickeners.
  Interventions: Other: Starch-based Thickened Liquids; Other: Xanthan-gum Thickened Liquids

INTERVENTIONS:
Other: Starch-based Thickened Liquids — Barium will be thickened to slightly, mildly, moderately and extremely thick consistences as defined by the International Dysphagia Diet Standardisation Initiative flow test.
  Other Names: Nestle Resource ThickenUp
Other: Xanthan-gum Thickened Liquids — Barium will be thickened to slightly, mildly, moderately and extremely thick consistences as defined by the International Dysphagia Diet Standardisation Initiative flow test.
  Other Names: Nestle Resource ThickenUp Clear

SUMMARY:
This study is part of a larger grant, for which the overall goal is to collect measurements of liquid flow through the oropharynx (i.e., mouth and throat) during swallowing. The focus of this study is to evaluate the flow of liquids of varying consistency in the head and neck cancer population.

DETAILED DESCRIPTION:
Thickened liquids are commonly used as an intervention for dysphagia (swallowing impairment). However, the field lacks a clear understanding of how liquids of different consistencies behave during swallowing. In order to improve understanding of the effectiveness of altered liquid consistency for improving dysphagia, the investigators are studying liquid flow through the oropharynx.

This study explores this question in individuals who have undergone radiation treatment for head and neck cancer, specifically located in the oropharynx.

Participants will swallow 20% w/v barium thickened to different consistencies (thin, slightly thick, and mildly thick) using commercially available food thickeners. Swallowing will be observed under videofluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* An initial cancer diagnosis of cancer in the base of tongue region of the oropharynx (Tumor staging T2,T3 & T4; Nodal staging N0 orN1; Human Papilloma Virus + or -).
* Completion of bilateral radiation therapy to the neck 3 months prior to enrollment
* No longer requiring primary enteral feeding for nutrition.

Exclusion Criteria:

* Prior history of swallowing, motor speech, gastro#esophageal difficulties, chronic sinusitis or taste disturbance.
* Previous radiation to the head and neck (prior to current illness);
* Previous cancer diagnosis;
* Prior or planned neck dissection;
* Trachestomy in situ;
* Neurological difficulties unrelated to spinal disorder (e.g. Stroke, Parkinson disease, etc).
* Cognitive communication difficulties that may hinder ability to participate.
* Current use of mechanical ventilation
* Type 1 Diabetes (due to the requirement to swallow stimuli containing starch based thickeners, which carry a significant carbohydrate load).
* Known allergies to latex, food coloring or dental glue (due to the probability that these items will come into contact with the oral mucosa during data collection).
* Occupational exposure to radiation exceeding 10 mSv in the past 6 months.
* Current pregnancy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who have recently completed radiation treatment for oropharynx cancer at the University Health Network, Toronto.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Steele, PhD, Principal Investigator — KITE - Toronto Rehabilitation Institute, University Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults With Oropharyngeal Cancer: Adult participants who had completed radiation therapy for oropharyngeal cancer within the past 3 months who underwent a swallowing x-ray study in which they swallowed liquid stimuli prepared to different consistencies.
Period: Overall Study
Arm/Group | Adults With Oropharyngeal Cancer
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adults With Oropharyngeal Cancer: Adult participants who have completed radiation therapy for oropharyngeal cancer within the past 3 months.
Arm/Group | Adults With Oropharyngeal Cancer
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 63 [49 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unsafe Swallowing
Description: Swallowing safety was measured using the Penetration-Aspiration Scale, an 8-point categorical scale which captures the depth to which any material enters the airway and whether or not the material is ejected. Levels 1 and 2 on the scale are considered safe, while levels > 2 are considered unsafe. Actual scale scores (1-8) will be recorded and then converted to binary categorical scores (< 3 vs >/= 3). We will report the frequency (count) of participants showing scores > 2 by bolus consistency.
Time Frame: Baseline (single timepoint only)
Population: Adult participants who had completed radiation therapy for oropharyngeal cancer within the past 3 months. A sample of 12 adults was enrolled. The thickened consistencies were only administered (and analyzed) for the 6 participants who displayed obvious unsafe swallowing on the thin liquid stimuli during data collection. A further 3 participants were determined to have shown unsafe swallowing on thin liquids during post-hoc analysis, but this was not recognized at the time of data collection.
Measure: Count of Participants; unit: Participants
Groups:
- Thin Liquid Barium: Participants were asked to take a series of 3 comfortable sips of thin liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder and water.
- Slightly Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of slightly thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, water and Nestle Resource ThickenUp Clear thickener.
- Mildly Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of mildly thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque barium powder, water and Nestle Resource ThickenUp Clear thickener.
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium
Number analyzed (Participants) | 12 | 6 | 6
Participants | 9 | 4 | 3

2. Primary Outcome: Amount of Residue in the Pharynx
Description: Residue is material remaining behind in the pharynx after the swallow. We measured residue by tracing the area of barium visible on a lateral view x-ray (in pixels, using ImageJ software) and dividing that area by the squared length C2-C4 cervical spine. This cervical spine scalar provides a common anatomical reference that is a proxy for pharyngeal size, and enables the comparison of residue severity across different people with different neck length and pharynx size. In healthy swallowing, residue is expected to be minimal. We report mean values and standard deviations for amount of residue by consistency (thin, slightly thick, and mildly thick liquids).
Time Frame: Baseline (single timepoint only)
Population: Adult participants who had completed radiation therapy for oropharyngeal cancer within the past 3 months. A sample of 12 adults was enrolled. The thickened consistencies were only administered (and analyzed) for the 6 participants who displayed unsafe swallowing on the thin liquid stimuli.
Measure: Mean (Standard Deviation); unit: % of the squared C2-C4 length scalar
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium
Number analyzed (Participants) | 12 | 6 | 6
% of the squared C2-C4 length scalar | 2.5 (2.7) | 3.3 (2.8) | 4.2 (3.1)

3. Secondary Outcome: Number of Participants Reporting Dislike of Thickened Liquid Stimuli
Description: Participants rated the palatability of lemon flavored water and liquid barium stimuli in slightly thick, mildly thick and moderately thick consistencies. Palatability was scored using a 9-point hedonic categorical rating system previously described by Pelletier et al. The ratings use 9 descriptors to capture the degree to which a participant likes a stimulus, with anchors of "Dislike extremely" and "Like extremely". Scores of 1-4 indicate liking of a stimulus, a score of 5 is neutral while scores of 6-9 indicate dislike. We dichotomized this scale between scores of 1-4 (liking) and scores of 5-9 and report the number of participants reporting scores of 6-9 (dislike).
Time Frame: Baseline (single timepoint only)
Population: Adult participants who had completed radiation therapy for oropharyngeal cancer within the past 3 months. A sample of 12 participants was enrolled. However, only 7 participants completed the palatability testing component of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Slightly Thick Lemon Flavored Water: Lemon flavored water mixed with Nestle Resource ThickenUp clear thickener to a slightly thick consistency.
- Slightly Thick Liquid Barium: Bracco E-Z-Paque barium prepared in 20% w/v concentration and mixed with water and Nestle Resource ThickenUp Clear thickener to a slightly thick consistency.
- Mildly Thick Lemon Flavored Water: Lemon flavored water mixed with Nestle Resource ThickenUp clear thickener to a mildly thick consistency.
- Mildly Thick Liquid Barium: Bracco E-Z-Paque barium prepared in 20% w/v concentration and mixed with water and Nestle Resource ThickenUp Clear thickener to a mildly thick consistency.
- Moderately Thick Lemon Flavored Water: Lemon flavored water mixed with Nestle Resource ThickenUp clear thickener to a moderately thick consistency.
Arm/Group | Slightly Thick Lemon Flavored Water | Slightly Thick Liquid Barium | Mildly Thick Lemon Flavored Water | Mildly Thick Liquid Barium | Moderately Thick Lemon Flavored Water
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
Participants | 2 | 3 | 3 | 5 | 4

ADVERSE EVENTS:
Time Frame: 1 week post data collection
Description: Participants experiencing any discomfort during or after participating in data collection were asked to report these to the study team. These were then reviewed for relatedness and seriousness.
Groups:
- Adults With Oropharyngeal Cancer: Adult participants who have completed radiation therapy for oropharyngeal cancer within the past 3 months will undergo a swallowing x-ray study in which they will swallow liquid stimuli prepared to different consistencies.
Arm/Group | Adults With Oropharyngeal Cancer
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04112940/Prot_SAP_000.pdf